CLINICAL TRIAL: NCT03918135
Title: Comparison of the Efficacy of Intravenous Paracetamol and Ibuprofen in Patients With Upper Respiratory Tract Infections Presenting With Fever in the Emergency Department
Brief Title: Comparison of the Efficacy of Intravenous Paracetamol and Ibuprofen in the Treatment of Fever Due to Upper Respiratory Tract Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Üzeyir Çimen, Research asistant, Pamukkale University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019TIPF002
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Fever
Keywords: fever, emergency department, paracetamol, ibuprofen, upper respiratory infection
MeSH Terms: conditions — Fever; Emergencies; Respiratory Tract Infections | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): Paracetamol 1000 mg of paracetamol (parol 10mg/ml solution Mefar,Turkey ) intravenous (IV) was given 100 patients
  Interventions: Drug: Paracetamol
- İbuprofen (Experimental): İbuprofen 400mg of ibuprofen (intrafen 400mg/4ml solution Gen ilaç sanayi,Turkey ) intravenous (IV) was given 100 patients
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Paracetamol — 1000 mg of paracetamol (parol 10mg/ml Mefar, Turkey) intravenous (IV) was given 100 patients
  Other Names:
  * Perfalgan
  * Paracerol
  Arms: Paracetamol
Drug: Ibuprofen — 400mg of ibuprofen(intrafen 400mg/4ml Gen ilaç sanayi, Turkey) intravenous (IV) was given 100 patients
  Other Names:
  Dorifen
  Arms: İbuprofen

SUMMARY:
Currently, paracetamol, ibuprofen and nonsteroidal antiinflammatory drugs are widely used by emergency physicians in Turkey for the treatment of fever . The objective of the study is compare the efficacy of intravenous ibuprofen and paracetamol in the treatment of patients with upper respiratory tract infections presenting with fever in the emergency department

DETAILED DESCRIPTION:
This is the randomized double blinded clinical trial to compare the efficacy of these two drugs in this clinical setting. A randomized clinical trial was conducted in the Emergency Department (ED) of Pamukkale University Medical Faculty Hospital Study personnel (emergency physicians and emergency service nurses) were trained before the study. When intravenous drugs (Paracetamol and İbuprofen) was being recommended, an eligibility checklist was completed by the attending physician. patients who presented to the emergency department with upper respiratory tract infection and had a temperature above 38.0 ° C were measured by a fever gauge included into the study First Group: 1000 mg of paracetamol ( parol 10mg/ml solution Mefar, Turkey) intravenous (IV) was given 100 patients

Second Group:

Ibuprofen 400 mg ( intrafen 400mg/4ml solution -Gen ilaç san., Turkey) intravenous (IV) was given 100 patients which determined to be applied as a group. Drug packs prepared in 150 ml serum physiology were numbered by an independent nurse, who not involved in the study Randomization was achieved by using computer software to generate random numbers. During the intervention, participants were monitored by an oxygen saturation (SpO2) monitor, an automatic sphygmomanometer (blood pressure), and a rhythm monitor (heart rate and rhythms). Patients in both groups received two types of medication in a similarmanner, thus ensuring double blind.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have fever for less than five days
* At least 1 upper respiratory tract infection (URTI) symptom according URTI questionare

Exclusion Criteria:

* Patients use anti-pyretic last 4 hours
* To be Pregnancy and breast-feeding Patients of childbearing age who are not using a birth control method
* Patients with an allergy trait (paracetamol and Ibuprofen) Illiterates
* Hemodynamically unstable patients
* Patients with renal transplantation
* Patients with glucose 6 phosphate dehydrogenase (G6PD) deficiency
* Patients with non-controlled hypertension
* Patients with a history of cerebrovascular disease
* Patients with severe liver, kidney,pulmonary and cardiac heart failure
* Patients use antibiotics last 7 days
* Patients with Wolff-Parkinson-White syndrome or accompanying arrhythmias associated with conductive stimulus delivery in the heart
* Patients with vision problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Decreasing of fever | Baseline and 120 minutes
  Comparison of the change of fever between the two groups. - (First group Paracetamol, Second Ibuprofen)

CONTACTS AND LOCATIONS:
Overall Officials: Atakan Yilmaz, MD, Principal Investigator — Pamukkale University; Gizem Oncel, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No